CLINICAL TRIAL: NCT02520310
Title: A Prospective, Multi-Center, Single-Arm Clinical Evaluation of the AVJ-514 System for the Treatment of Symptomatic Chronic Severe Mitral Regurgitation
Brief Title: AVJ-514 Japan Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVJ-514
Record Dates: First submitted 2015-07-17; First posted 2015-08-11 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Mitral Stenosis With Insufficiency; Functional Mitral Regurgitation; Mitral Insufficiency; Mitral Valve Incompetence; Mitral Valve Regurgitation
Keywords: Mitral Regurgitation; mitral valve surgery; AVJ-514 Delivery System; Symptomatic Heart Failure; Heart Valve Disease
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AVJ-514 (Experimental): The AVJ-514 system
  Interventions: Device: AVJ-514

INTERVENTIONS:
Device: AVJ-514 — Patients receiving AVJ-514 device

SUMMARY:
The objective of the study is to confirm the reproducibility of the evidence of safety and efficacy of AVJ-514 System technology in Japanese subjects who have been deemed difficult for mitral valve surgery by the local site heart team.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, single-arm clinical evaluation of the AVJ-514 System for the treatment of symptomatic chronic severe mitral regurgitation (MR) in Japanese subjects deemed difficult for mitral valve surgery by the local site heart team.

Patients will be evaluated at baseline, discharge, 30 days, 6 months, 1 year, 2 years, 3 years, 4 years, and 5 years in Japanese Medical Centers.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria:

1. Age 20 years or older.
2. Symptomatic moderate-to-severe (3+) or severe MR (4+) chronic Degenerative Mitral Regurgitation (DMR) or Functional Mitral Regurgitation (FMR) determined by assessment of a qualifying transthoracic echocardiogram (TTE) obtained within 90 days and transesophageal echocardiogram (TEE) obtained within180 days prior to subject registration, with MR severity based principally on the TTE study and confirmed by the Echocardiography Core Laboratory (ECL). The ECL may request a TEE.
3. Left Ventricular Ejection Fraction (LVEF) is ≥ 30％ within 90 days prior to subject registration, assessed by the site using any one of the following methods: echocardiography, contrast left ventriculography, gated blood pool scan or cardiac magnetic resonance imaging (MRI). Note: The method must provide a quantitative readout (not a visual assessment).
4. New York Heart Association (NYHA) classification is class II, class III, or ambulatory class IV.
5. Subject is deemed difficult for mitral valve surgery due to either Society of Thoracic Surgery (STS) surgical mortality risk for mitral valve replacement of ≥ 8% OR due to the presence of one of the following risk factors:

   * Porcelain aorta or mobile ascending aortic atheroma
   * Post-radiation mediastinum
   * Previous mediastinitis
   * Functional MR with LVEF < 40%
   * Over 75 years old with LVEF < 40%
   * Re-operation with patent grafts
   * Two or more prior cardiothoracic surgeries
   * Hepatic cirrhosis
   * Other surgical risk factor(s)
6. Mitral valve area ≥ 4.0 cm2 assessed by ECL based TTE within 90 days prior to subject registration. The ECL may request a TEE.
7. Left Ventricular End Systolic Dimension (LVESD) is ≤ 60mm assessed by site based on the TTE obtained within 90 days prior to subject registration.
8. The primary regurgitant jet is non-commissural based on TEE, and in the opinion of the AVJ-514 implanting investigator can successfully be treated by the AVJ-514. If a secondary jet exists, it must be considered clinically insignificant.
9. Transseptal catheterization and femoral vein access is determined to be feasible by the treating physician.
10. The subject or the subject's legal representative has been informed of the nature of the study and agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board of the respective clinical site.

Exclusion Criteria:

Subjects must not meet any of the following exclusion criteria:

1. LVEF is < 30%
2. Leaflet anatomy which may preclude AVJ-514 implantation, proper positioning on the leaflets or sufficient reduction in MR by the AVJ-514 based. This evaluation is based on TEE evaluation of the mitral valve within 180 days prior to subject registration and includes:

   * Insufficient mobile leaflet available for grasping with the AVJ-514 device
   * Lack of both primary and secondary chordal support in the grasping area
   * Evidence of significant calcification in the grasping area
   * Presence of a significant cleft in the grasping area
3. Life expectancy < 1 year due to associated non-cardiac co-morbid conditions
4. Need for emergent or urgent surgery for any reason
5. Prior open heart mitral valve leaflet surgery or any currently implanted prosthetic mitral valve or any prior transcatheter mitral valve procedure.
6. Echocardiographic evidence of intracardiac mass, thrombus or vegetation.
7. Active endocarditis or active rheumatic heart disease or leaflets degenerated from rheumatic disease (i.e. noncompliant, perforated).
8. Untreated clinically significant coronary artery disease requiring revascularization or significant myocardial ischemia or evidence of an acute myocardial infarction in the prior 90 days of registration.
9. Cerebrovascular accident within 180 days prior to registration
10. Severe symptomatic carotid stenosis (> 70% by ultrasound)
11. Any cardiac surgery within 180 days prior to registration
12. Percutaneous coronary intervention (PCI) within the last 30 days prior to registration
13. Implant of Cardiac Resynchronization Therapy (CRT), Cardiac Resynchronization Therapy with Cardioverter Defibrillator (CRT-D) pacemaker or Implantable Cardioverter Defibrillator (ICD)within the last 30 days prior to registration.
14. Transcatheter aortic valve replacement (TAVR) within the last 30 days prior to registration.
15. Severe tricuspid regurgitation or aortic valve disease requiring surgical treatment.
16. In the judgment of the Investigator, the femoral vein cannot accommodate a 24 F catheter or presence of ipsilateral deep vein thrombosis (DVT).
17. Hemodynamic instability defined as systolic pressure < 90 mmHg without afterload reduction drug or cardiogenic shock or intra-aortic balloon pump.
18. History of bleeding diathesis or coagulopathy or subject will refuse blood transfusions.
19. Active infections requiring current antibiotic therapy (if temporary illness, patients may enroll at least 14 days after discontinuation of antibiotics). Patients must be free from infection prior to treatment. Any required dental work should be completed a minimum of 21 days prior to treatment.
20. Intravenous drug abuse or suspected inability to adhere to follow-up.
21. Patients in whom TEE is contraindicated.
22. A known hypersensitivity or contraindication to study or procedure medications which cannot be adequately managed medically.
23. In the judgment of the Investigator, subjects in whom the presence of a permanent pacemaker or pacing leads would interfere with placement of the test device or the placement of the test device would disrupt the leads.
24. Subject intends to participate in any other investigational or invasive clinical study within a period of 1 year following the AVJ-514 procedure.
25. Currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the current study endpoints. (Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials).
26. In the opinion of the investigator or designee, subject is unable to comply with the requirements of the study protocol or is unsuitable for the study for any reason.
27. In the opinion of the anesthesiologist, general anesthesia is contraindicated.
28. Pregnant or planning pregnancy within next 1 year.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-09-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2021-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryohei Yozu, MD, PhD, Principal Investigator — Keio University; Morimasa Takayama, MD, PhD, Principal Investigator — Sakakibara Heart Institute; Peter Staehr, MD, Study Director — Abbott Vascular, Inc.
Locations (6):
- Japan (6):
  - Shonan Kamakura General Hospital, Kanagawa
  - Sendai Kosei Hospital, Miyagi
  - National Cerebral and Cardiovascular Center, Osaka
  - Keio University Hospital, Tokyo
  - Sakakibara Heart Institute, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo

REFERENCES:
- [Derived] Hayashida K, Yasuda S, Matsumoto T, Amaki M, Mizuno S, Tobaru T, Jujo K, Ootomo T, Yamaguchi J, Fukuda K, Saito S, Foster E, Qasim A, Kitakaze M, Yozu R, Takayama M. AVJ-514 Trial - Baseline Characteristics and 30-Day Outcomes Following MitraClip(R) Treatment in a Japanese Cohort. Circ J. 2017 Jul 25;81(8):1116-1122. doi: 10.1253/circj.CJ-17-0115. Epub 2017 Mar 17. PMID 28321004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 subjects were enrolled at 6 japan sites from September 7, 2015 to June 14, 2016.
Pre-assignment Details: Prior to the procedure,subjects were assessed to ensure there was no significant change in the subject's overall condition (e.g.stroke,MI,active infection,etc.) that would preclude treatment. If the subject experienced any significant change, the subject was treated&reassessed for the clinical investigation.They were not considered registered.
Groups:
- AVJ-514: This study contains only one group. All patients received AVJ-514 device - MitraClip NT System.
Period: At 30 Days Clinical Follow-up
Arm/Group | AVJ-514
Started | 30
Completed | 30
Not Completed | 0
Period: At 6 Months Clinical Follow-up
Arm/Group | AVJ-514
Started | 30
Completed | 29
Not Completed | 1
Not completed — Death | 1
Period: At 1 Year Clinical Follow-up
Arm/Group | AVJ-514
Started | 29
Completed | 28
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: At 2 Year Clinical Follow-up
Arm/Group | AVJ-514
Started | 28
Completed | 28
Not Completed | 0
Period: AT 3 Year Clinical Follow-up
Arm/Group | AVJ-514
Started | 28
Completed | 24
Not Completed | 4
Not completed — Death | 2
Not completed — Withdrawal by Subject | 2
Period: AT 4 Year Clinical Follow-up
Arm/Group | AVJ-514
Started | 24
Completed | 22
Not Completed | 2
Not completed — Death | 1
Not completed — missed visit | 1

BASELINE CHARACTERISTICS:
Groups:
- AVJ-514: The AVJ-514 system: Patients receiving AVJ-514 device
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Procedure Success (APS)
Description: APS is defined as successful implantation of the AVJ-514 device(s) with resulting MR severity of 2+ or less as determined by the Echocardiographic Core Laboratory (ECL) assessment of a discharge echocardiogram. Subjects who die or who undergo mitral valve surgery before discharge are an APS failure.
Time Frame: On day 0 (the day of procedure)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 26

2. Secondary Outcome: Percentage of Participants With Major Adverse Events (MAE) at 30 Days
Description: MAE is a composite of death, stroke, myocardial infarction (MI), renal failure, and non-elective cardiovascular surgery for device or procedure related adverse events occurring after the femoral vein puncture for transseptal access. This outcome measure calculates the percentage of participants with MAE at 30 days (= total subjects with MAE/total subjects enrolled).
Time Frame: 30 days
Population: Intention-to-Treat (ITT) population is defined as all the subjects who have registered in the study and have AVJ-514 clip device placement attempted.
Measure: Number; unit: percentage of participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
percentage of participants
  Death | 0
  Stroke | 0
  Myocardial infarction | 0
  Renal failure | 0
  Procedure related adverse events | 0

3. Secondary Outcome: Percentage of Participants With MAE at 1 Year
Description: as for outcome 2
Time Frame: 1 year
Population: ITT population is defined as all the subjects who have registered in the study and have AVJ-514 clip device placement attempted. This section talks about MAE at 1 year. A total of two MAES were reported through 1 year. 1 MAE for Death and 1 MAE for Renal Failure.
Measure: Number; unit: percentage of participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
percentage of participants
  Death | 3.3
  Stroke | 0
  Myocardial infarction | 0
  Renal failure | 3.3
  Procedure related adverse events | 0

4. Secondary Outcome: Number of Participants With MAE Occurring After the Femoral Vein Puncture for Transseptal Access
Description: MAE listed below will be adjudicated by the Clinical Events Committee at 30 days:
  * Death
  * Stroke
  * Myocardial infarction
  * Renal failure
  * Non-elective cardiovascular surgery for device or procedure related adverse events
Time Frame: 30 days
Population: ITT population is defined as all the subjects who have registered in the study and have AVJ-514 clip device placement attempted.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

5. Secondary Outcome: Number of Participants With Mitral Valve Stenosis Requiring Surgery
Description: Defined as a mitral valve orifice of less than 1.5 cm^2 as measured by the Echocardiography Core Laboratory.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

6. Secondary Outcome: Number of Participants With Mitral Valve Stenosis Not Requiring Surgery
Description: Defined as a mitral valve orifice of less than 1.5 cm^2 as measured by the Echocardiography Core Laboratory.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

7. Secondary Outcome: Number of Participants With Single Leaflet Device Attachment (SLDA) Requiring Surgery
Description: SLDA is defined as attachment of one mitral valve leaflet to the AVJ-514 device.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

8. Secondary Outcome: Number of Participants With Single Leaflet Device Attachment (SLDA) Not Requiring Surgery
Description: SLDA is defined as attachment of one mitral valve leaflet to the AVJ-514 device.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 1

9. Secondary Outcome: Number of Participants With Iatrogenic Atrial Septal Defect
Description: Defined as defect ('hole') in the septum between the left and right atria; considered clinically significant if it requires percutaneous or surgical intervention.
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

10. Secondary Outcome: Percentage of Participants With Device Implant Rate
Description: Defined as the rate of successful delivery and deployment of one or more AVJ-514 device with echocardiographic evidence of leaflet approximation and retrieval of the delivery catheter.
Time Frame: On the day of procedure
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
percentage of participants
  0 | 0
  1 | 30
  2 | 63
  >=3 | 7

11. Secondary Outcome: Device Procedure Time
Description: Defined as the time elapsed from the start of the transseptal procedure to the time the Steerable Guide Catheter is removed.
Time Frame: On the day of procedure
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Minutes | 206.4 (84.06)

12. Secondary Outcome: Total Procedure Time
Description: Defined as the time elapsed from the first of any of the following: intravascular catheter placement, anesthesia or sedation, or transesophageal echocardiogram (TEE), to the removal of the last catheter and TEE.
Time Frame: On the day of procedure
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Minutes | 284.6 (90.67)

13. Secondary Outcome: Device Time
Description: Defined as the time the Steerable Guide Catheter is placed in the intra-atrial septum until the time the AVJ-514 Delivery System (CDS) is retracted into the Steerable Guide Catheter.
Time Frame: On the day of procedure
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Minutes | 126.6 (79.57)

14. Secondary Outcome: Fluoroscopy Duration
Description: Defined as the duration of exposure to fluoroscopy during the AVJ-514 procedure.
Time Frame: On the day of procedure
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Minutes | 62.5 (31.11)

15. Secondary Outcome: Length of Stay in Intensive Care Unit (ICU)/Critical Care Unit (CCU)/Post-Anesthesia Care Unit (PACU) (ICU/CCU/PACU)
Description: Length of stay in ICU/CCU/PACU is cumulative hours of Hospital stay in (PACU/CCU/ICU)
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
Hours | 36.8 (36.31)

16. Secondary Outcome: Length of Hospital Stay Excluding Rehabilitation Stay
Description: Length of hospital stay excluding rehabilitation stay = Length of hospital stay (Date of Discharge - Date of Admission)
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Days | 14.4 (8.53)

17. Secondary Outcome: Length of Rehabilitation Stay
Description: Cumulative days of rehabilitation stay during hospitalization.
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AVJ-514
Number analyzed (Participants) | 5
Days | 4.9 (3.12)

18. Secondary Outcome: Percentage of Participants With Discharge Status
Description: Location to which subject was discharged (home or another facility).
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
percentage of participants
  Released to home | 96.7
  Released to rehab facility or skilled nursing home | 3.3
  Returned to rehab facility or skilled nursing home | 0
  Transferred to another hospital | 0
  Subject died | 0
  Other | 0

19. Secondary Outcome: Length of Stay (Not at Baseline Facility)
Description: If subject discharged to another facility (different from baseline facility), length of stay at facility to which subject was discharged. Length of Stay (not at baseline facility) = Sum for all eligible log lines which had been entered in Electronic Data Capture (EDC) for ICU/CCU/PACU and rehabilitation.
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
Days | 2.6 (2.66)

20. Secondary Outcome: Number of Participants With Mitral Regurgitation (MR) Severity Grade
Description: Mitral regurgitation severity is determined based on the American Society of Echocardiography (ASE) Recommendations for Evaluation of The Severity of Native Valvular Regurgitation with Two-Dimensional and Doppler Echocardiography. MR severity grade was assessed by the core lab using the transthoracic echocardiogram (TTE) at baseline, discharge and subsequent follow-up visits. The severity of MR is determined by the amount of blood being pushed back into the left atrium when it should be circulating through the left ventricle with each heart beat. MR severity is typically classified as mild (grade 1+), moderate (grade 2+), moderate to severe (grade 3+) or severe (grade 4+).
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  MR Severity Grade 0 | 0
  MR Severity Grade 1+ | 0
  MR Severity Grade 2+ | 0
  MR Severity Grade 3+ | 24
  MR Severity Grade 4+ | 6

21. Secondary Outcome: Number of Participants With MR Severity Grade
Description: as for outcome 20
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  MR severity grade 0 | 0
  MR severity grade 1+ | 21
  MR severity grade 2+ | 5
  MR severity grade 3+ | 4
  MR severity grade 4+ | 0

22. Secondary Outcome: Number of Participants With MR Severity Grade
Description: as for outcome 20
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  MR severity grade 0 | 0
  MR severity grade 1+ | 17
  MR severity grade 2+ | 9
  MR severity grade 3+ | 4
  MR severity grade 4+ | 0

23. Secondary Outcome: Number of Participants With MR Severity Grade
Description: as for outcome 20
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
Participants
  MR severity grade 0 | 0
  MR severity grade 1+ | 14
  MR severity grade 2+ | 9
  MR severity grade 3+ | 6
  MR severity grade 4+ | 0

24. Secondary Outcome: Number of Participants With MR Severity Grade
Description: as for outcome 20
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
Participants
  MR severity grade 0 | 0
  MR severity grade 1+ | 8
  MR severity grade 2+ | 13
  MR severity grade 3+ | 7
  MR severity grade 4+ | 0

25. Secondary Outcome: MR Severity Grade
Description: as for outcome 20
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
Participants
  MR 0 | 0
  MR 1+ | 12
  MR 2 + | 13
  MR 3+ | 2
  MR 4+ | 1

26. Secondary Outcome: MR Severity Grade
Description: as for outcome 20
Time Frame: 3 years
Population: All subjects woth availble data
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
Participants
  MR 0+ | 0
  MR 1+ | 10
  MR 2+ | 10
  MR 3+ | 4
  MR 4 + | 0

27. Secondary Outcome: MR Severity Grade
Description: as for outcome 20
Time Frame: 4 years
Population: All available data is reported
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 22
Participants
  MR 0+ | 0
  MR 1+ | 7
  MR 2+ | 9
  MR 3+ | 5
  MR 4+ | 0
  Not Available | 1

28. Secondary Outcome: MR Severity Grade
Time Frame: 5 years
Reporting Status: Not Posted

29. Secondary Outcome: Regurgitant Volume (RV)
Description: Regurgitant volume as determined by the Echocardiographic Core Laboratory (ECL). In the presence of regurgitation of one valve, without any intracardiac shunt, the flow through the affected valve is larger than through other competent valves. The difference between the two represents the regurgitant volume.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
mL/beat | 29.5 (21.0)

30. Secondary Outcome: Regurgitant Volume (RV)
Description: as for outcome 29
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 17
mL/beat | 11.4 (9.5)

31. Secondary Outcome: Regurgitant Volume (RV)
Description: as for outcome 29
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 19
mL/beat | 16.9 (12.3)

32. Secondary Outcome: Regurgitant Volume (RV)
Description: as for outcome 29
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 22
mL/beat | 16.9 (15.0)

33. Secondary Outcome: Regurgitant Volume (RV)
Description: as for outcome 29
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 19
mL/beat | 15.1 (13.6)

34. Secondary Outcome: Regurgitant Volume (RV)
Description: Regurgitant volume as determined by the site. In the presence of regurgitation of one valve, without any intracardiac shunt, the flow through the affected valve is larger than through other competent valves. The difference between the two represents the regurgitant volume.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 15
ml/beat | 27.1 (18.9)

35. Secondary Outcome: Regurgitant Volume (RV)
Description: as for outcome 34
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 16
ml/beat | 36.5 (22.5)

36. Secondary Outcome: Regurgitant Volume (RV)
Description: as for outcome 34
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml/beat
Arm/Group | AVJ-514
Number analyzed (Participants) | 10
ml/beat | 44.0 (22.6)

37. Secondary Outcome: Regurgitant Volume (RV)
Time Frame: 5 years
Reporting Status: Not Posted

38. Secondary Outcome: Regurgitant Fraction (RF)
Description: Regurgitant fraction as determined by the Echocardiographic Core Laboratory (ECL). Regurgitant fraction is defined as the regurgitant volume divided by the forward stroke volume through the regurgitant valve.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
percentage of regurgitant fraction | 36 (16.1)

39. Secondary Outcome: Regurgitant Fraction (RF)
Description: as for outcome 38
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 17
percentage of regurgitant fraction | 18.7 (13.4)

40. Secondary Outcome: Regurgitant Fraction (RF)
Description: as for outcome 38
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 19
percentage of regurgitant fraction | 22.9 (14.4)

41. Secondary Outcome: Regurgitant Fraction (RF)
Description: as for outcome 38
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 22
percentage of regurgitant fraction | 23.9 (16.0)

42. Secondary Outcome: Regurgitant Fraction (RF)
Description: as for outcome 38
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 19
percentage of regurgitant fraction | 22.2 (15.3)

43. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: Left Ventricular End Diastolic Volume (LVEDV) as measured by the Echocardiography Core Laboratory (ECL). Left Ventricular end-diastolic volume (LVEDV) measured using 2-dimensional echocardiography. The endocardium is traced at end-diastole (frame before mitral valve closure or maximum cavity dimension) in the 2- and 4-chamber views to calculate volumes.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
mL | 144.1 (47.2)

44. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: as for outcome 43
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
mL | 126.4 (40.5)

45. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: as for outcome 43
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
mL | 130.0 (37.9)

46. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: Left Ventricular End Diastolic Volume (LVEDV) as measured by the Echocardiography Core Laboratory (ECL). Left Ventricular enddiastolic volume (LVEDV) measured using 2-dimensional echocardiography. The endocardium is traced at end-diastole (frame before mitral valve closure or maximum cavity dimension) in the 2- and 4-chamber views to calculate volumes.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
mL | 134.6 (40.7)

47. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: as for outcome 43
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
mL | 127.0 (43.4)

48. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: Left Ventricular End Diastolic Volume (LVEDV) as measured by the site. Left Ventricular enddiastolic volume (LVEDV) measured using 2-dimensional echocardiography. The endocardium is traced at end-diastole (frame before mitral valve closure or maximum cavity dimension) in the 2- and 4-chamber views to calculate volumes.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
ml | 147.3 (59.2)

49. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: as for outcome 48
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
ml | 144.6 (61.4)

50. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Description: as for outcome 48
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
ml | 138.9 (63.6)

51. Secondary Outcome: Left Ventricular End Diastolic Volume (LVEDV)
Time Frame: 5 years
Reporting Status: Not Posted

52. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: Left Ventricular End Systolic Volume (LVESV) as measured by the Echocardiography Core Laboratory (ECL). Left Ventricular end-systolic volume (LVESV) measured using 2-dimensional echocardiography. The endocardium is traced at end-systole (frame prior to mitral valve opening or the minimum cavity area) in the 2- and 4-chamber views to calculate volumes.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
mL | 74.1 (34.3)

53. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 52
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
ml | 72.6 (36.5)

54. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 52
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
mL | 68.7 (32.2)

55. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 52
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
mL | 72.5 (39.9)

56. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 52
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
mL | 69.5 (38.8)

57. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: Left Ventricular End Systolic Volume (LVESV) as measured by the site. Left Ventricular end-systolic volume (LVESV) measured using 2-dimensional echocardiography. The endocardium is traced at end-systole (frame prior to mitral valve opening or the minimum cavity area) in the 2- and 4-chamber views to calculate volumes.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
ml | 83.9 (51.9)

58. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 57
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
ml | 87.0 (53.3)

59. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Description: as for outcome 57
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
ml | 83.7 (57.3)

60. Secondary Outcome: Left Ventricular End Systolic Volume (LVESV)
Time Frame: 5 years
Reporting Status: Not Posted

61. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the Echocardiography Core Laboratory (ECL).
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
cm | 5.7 (0.9)

62. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the Echocardiography Core Laboratory (ECL).
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
cm | 5.4 (0.8)

63. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the Echocardiography Core Laboratory (ECL).
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
cm | 5.5 (0.8)

64. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the Echocardiography Core Laboratory (ECL).
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
cm | 5.6 (0.9)

65. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the Echocardiography Core Laboratory (ECL).
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
cm | 5.4 (0.8)

66. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the site.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
cm | 5.7 (0.9)

67. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the site.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
cm | 5.6 (1.0)

68. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Description: Left Ventricular End Diastolic Dimension (LVEDD) as measured by the site
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
cm | 5.7 (0.9)

69. Secondary Outcome: Left Ventricular End Diastolic Dimension (LVEDD)
Time Frame: 5 years
Reporting Status: Not Posted

70. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the ECL.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
cm | 4.1 (1.2)

71. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the ECL.
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
cm | 4.1 (1.1)

72. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the ECL.
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
cm | 4.1 (1.2)

73. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the ECL.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
cm | 4.1 (1.2)

74. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the ECL.
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
cm | 4.1 (1.1)

75. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the site.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
cm | 4.3 (1.2)

76. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the site.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
cm | 4.4 (1.3)

77. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Description: Left Ventricular End Systolic Dimension (LVESD) as measured by the site.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
cm | 4.4 (1.2)

78. Secondary Outcome: Left Ventricular End Systolic Dimension (LVESD)
Time Frame: 5 years
Reporting Status: Not Posted

79. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as measured by the ECL.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
percentage of ejection fraction | 50.2 (12.8)

80. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as measured by the ECL.
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
percentage of ejection fraction | 45.0 (11.8)

81. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as measured by the ECL.
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
percentage of ejection fraction | 49.8 (12.6)

82. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as measured by the ECL.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
percentage of ejection fraction | 49.5 (15.2)

83. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as measured by the ECL.
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
percentage of ejection fraction | 48.7 (14.2)

84. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as measured by the site.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
percentage of ejection fraction | 47.0 (15.1)

85. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Description: Left Ventricular Ejection Fraction (LVEF) as measured by the site.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
percentage of ejection fraction | 44.8 (15.9)

86. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of Ejection Fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
percentage of Ejection Fraction | 44.5 (17.8)

87. Secondary Outcome: Left Ventricular Ejection Fraction (LVEF)
Time Frame: 5 years
Reporting Status: Not Posted

88. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: Pulmonary Artery Systolic Pressure (PASP) is presented in place of Right Ventricular Systolic Pressure (RVSP). PASP is equal to RVSP in the absence of pulmonic stenosis.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
mmHg | 40.2 (13.0)

89. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 20
mmHg | 35.1 (5.5)

90. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 20
mmHg | 37.3 (8.6)

91. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 22
mmHg | 35.4 (8.6)

92. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 23
mmHg | 35.3 (10.9)

93. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: 24 months
Reporting Status: Not Posted

94. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: 3 years
Reporting Status: Not Posted

95. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: 4 years
Reporting Status: Not Posted

96. Secondary Outcome: Pulmonary Artery Systolic Pressure (PASP)
Description: as for outcome 88
Time Frame: 5 years
Reporting Status: Not Posted

97. Secondary Outcome: Mitral Valve Area (MVA)
Description: It is the orifice area of the mitral valve.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
cm^2 | 6.0 (1.1)

98. Secondary Outcome: Mitral Valve Area (MVA)
Description: It is the orifice area of the mitral valve.
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
cm^2 | 2.8 (0.6)

99. Secondary Outcome: Mitral Valve Area (MVA)
Description: It is the orifice area of the mitral valve.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 26
cm^2 | 2.8 (0.8)

100. Secondary Outcome: Mitral Valve Area(MVA)
Description: It is the orifice area of the mitral valve.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 26
cm^2 | 2.3 (0.6)

101. Secondary Outcome: Mitral Valve Area(MVA)
Description: It is the orifice area of the mitral valve.
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 23
cm^2 | 2.4 (0.6)

102. Secondary Outcome: Mitral Valve Area (MVA)
Description: It is the orifice area of the Mitral Valve
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 26
cm^2 | 2.9 (0.8)

103. Secondary Outcome: Mitral Valve Area (MVA)
Description: It is the orifice area of the Mitral Valve.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 20
cm^2 | 3.6 (1.9)

104. Secondary Outcome: Mitral Valve Area (MVA)
Description: It is the orifice area of the Mitral Valve.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: cm^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 17
cm^2 | 2.9 (0.7)

105. Secondary Outcome: Mitral Valve Area (MVA)
Time Frame: 5 years
Reporting Status: Not Posted

106. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by the Echocardiography Core Laboratory (ECL).
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
mmHg | 2.4 (0.7)

107. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: as for outcome 106
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 27
mmHg | 3.6 (2.0)

108. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: as for outcome 106
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
mmHg | 3.7 (1.8)

109. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: as for outcome 106
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 23
mmHg | 4.1 (2.2)

110. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: as for outcome 106
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
mmHg | 3.8 (1.2)

111. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by the site.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
mmHg | 3.0 (1.4)

112. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by the site.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
mmHg | 3.6 (1.5)

113. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Description: Defined as the mean and peak pressure gradients across the mitral valve as measured by the site.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
mmHg | 3.6 (1.3)

114. Secondary Outcome: Mean Mitral Valve Pressure Gradient (MVG)
Time Frame: 5 years
Reporting Status: Not Posted

115. Secondary Outcome: Number of Participants With Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the ECL.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Yes | 0
  No | 29
  Not evaluable | 1

116. Secondary Outcome: Number of Participants With Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the ECL
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Yes | 0
  No | 30
  Not evaluable | 0

117. Secondary Outcome: Number of Participants With Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the ECL
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Yes | 0
  No | 30
  Not evaluable | 0

118. Secondary Outcome: Number of Participants With Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the ECL
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
Participants
  Yes | 1
  No | 28
  Not evaluable | 0

119. Secondary Outcome: Number of Participants With Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the ECL
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
Participants
  Yes | 0
  No | 28
  Not evaluable | 0

120. Secondary Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the site.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
Participants
  Yes | 0
  No | 28
  Not Evaluable | 0

121. Secondary Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the site.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
Participants
  Yes | 0
  No | 24
  Not Evaluable | 0

122. Secondary Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Description: Systolic Anterior Motion (SAM) of the mitral valve is measured by the site.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 22
Participants
  Yes | 0
  No | 21
  Not Evaluable | 1

123. Secondary Outcome: Systolic Anterior Motion of the Mitral Valve (Present or Absent)
Time Frame: 5 years
Reporting Status: Not Posted

124. Secondary Outcome: Forward Stroke Volume (FSV)
Description: Defined as the volume of blood pumped from the left ventricle per heartbeat.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
ml | 46.8 (12.3)

125. Secondary Outcome: Forward Stroke Volume (FSV)
Description: Defined as the volume of blood pumped from the left ventricle per heartbeat.
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
ml | 52.6 (14.7)

126. Secondary Outcome: Forward Stroke Volume (FSV)
Description: Defined as the volume of blood pumped from the left ventricle per heartbeat.
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
ml | 56.4 (12.9)

127. Secondary Outcome: Forward Stroke Volume (FSV)
Description: Defined as the volume of blood pumped from the left ventricle per heartbeat.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
ml | 49.2 (9.6)

128. Secondary Outcome: Forward Stroke Volume (FSV)
Description: Defined as the volume of blood pumped from the left ventricle per heartbeat.
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
ml | 49.6 (13.8)

129. Secondary Outcome: Forward Stroke Volume (FSV)
Time Frame: 24 months
Reporting Status: Not Posted

130. Secondary Outcome: Forward Stroke Volume (FSV)
Time Frame: 3 years
Reporting Status: Not Posted

131. Secondary Outcome: Forward Stroke Volume (FSV)
Time Frame: 4 years
Reporting Status: Not Posted

132. Secondary Outcome: Forward Stroke Volume (FSV)
Time Frame: 5 years
Reporting Status: Not Posted

133. Secondary Outcome: Cardiac Output (CO)
Description: Cardiac output as measured by the Echocardiographic Core Laboratory (ECL). Cardiac output is the product of forward stroke volume and heart rate.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
L/min | 3.0 (0.7)

134. Secondary Outcome: Cardiac Output (CO)
Description: as for outcome 133
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
L/min | 3.1 (0.8)

135. Secondary Outcome: Cardiac Output (CO)
Description: as for outcome 133
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
L/min | 3.5 (1.1)

136. Secondary Outcome: Cardiac Output (CO)
Description: as for outcome 133
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
L/min | 3.1 (0.7)

137. Secondary Outcome: Cardiac Output (CO)
Description: as for outcome 133
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
L/min | 3.2 (1.2)

138. Secondary Outcome: Cardiac Output (CO)
Description: Cardiac output as measured by the site. Cardiac output is the product of forward stroke volume and heart rate.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 27
L/min | 4.1 (1.8)

139. Secondary Outcome: Cardiac Output (CO)
Description: Cardiac output as measured by the site. Cardiac output is the product of forward stroke volume and heart rate.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
L/min | 5.6 (8.9)

140. Secondary Outcome: Cardiac Output (CO)
Description: Cardiac output as measured by the site. Cardiac output is the product of forward stroke volume and heart rate.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
L/min | 6.3 (9.3)

141. Secondary Outcome: Cardiac Output (CO)
Time Frame: 5 years
Reporting Status: Not Posted

142. Secondary Outcome: Cardiac Index (CI)
Description: Cardiac index is defined as cardiac output divided by body surface area. Cardiac Index was measured by the Echocardiographic Core Laboratory (ECL).
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
L/min/m^2 | 2 (0.4)

143. Secondary Outcome: Cardiac Index (CI)
Description: as for outcome 142
Time Frame: At Discharge (≤ 14.4 ± 8.5 days post index procedure)
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
L/min/m^2 | 2.1 (0.6)

144. Secondary Outcome: Cardiac Index (CI)
Description: as for outcome 142
Time Frame: 30 days
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
L/min/m^2 | 2.3 (0.8)

145. Secondary Outcome: Cardiac Index (CI)
Description: as for outcome 142
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
L/min/m^2 | 2.0 (0.5)

146. Secondary Outcome: Cardiac Index (CI)
Description: as for outcome 142
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
L/min/m^2 | 2.1 (0.7)

147. Secondary Outcome: Cardiac Index (CI)
Description: Cardiac index is defined as cardiac output divided by body surface area. Cardiac Index was measured by the site.
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 27
L/min/m^2 | 2.6 (1.1)

148. Secondary Outcome: Cardiac Index (CI)
Description: Cardiac index is defined as cardiac output divided by body surface area. Cardiac Index was measured by the site.
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
L/min/m^2 | 3.6 (5.7)

149. Secondary Outcome: Cardiac Index (CI)
Description: Cardiac index is defined as cardiac output divided by body surface area. Cardiac Index was measured by the site.
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: L/min/m^2
Arm/Group | AVJ-514
Number analyzed (Participants) | 19
L/min/m^2 | 4.1 (5.5)

150. Secondary Outcome: Cardiac Index (CI)
Time Frame: 5 years
Reporting Status: Not Posted

151. Secondary Outcome: Number of Participants With All-cause Mortality
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 1

152. Secondary Outcome: All-cause Mortality
Time Frame: 24 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 1

153. Secondary Outcome: All-cause Mortality
Time Frame: 3 years
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

154. Secondary Outcome: All-cause Mortality
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 5

155. Secondary Outcome: All-cause Mortality
Time Frame: 5 years
Reporting Status: Not Posted

156. Secondary Outcome: Number of Participants With the Primary Safety Composite of MAE at 1 Year
Description: MAE is a composite of death, stroke, MI, renal failure, and non-elective cardiovascular surgery for device or procedure related adverse events occurring after the femoral vein puncture for transseptal access. No of Participants with the MAEs at 12 months. One death and One Renal Failure was reported in two subjects.
Time Frame: 12 months
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Death | 1
  Stroke | 0
  MI | 0
  Renal failure | 1
  Non-elective cardiovascular surgery | 0

157. Secondary Outcome: Freedom From the Components of the Primary Safety Composite of MAE
Description: MAE is a composite of death, stroke, MI, renal failure, and non-elective cardiovascular surgery for device or procedure related adverse events occurring after the femoral vein puncture for transseptal access.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Death | 1
  Stroke | 1
  Myocardial Infarction | 0
  Renal Failure | 1
  Non-Elective Cardiovascular Sugery | 0

158. Secondary Outcome: Freedom From the Components of the Primary Safety Composite of MAE
Description: as for outcome 157
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Death | 3
  Stroke | 1
  Myocardial Infarction | 0
  Renal Failure | 2
  Non-elective cardiovascular surgery | 0

159. Secondary Outcome: Freedom From the Components of the Primary Safety Composite of MAE
Description: as for outcome 157
Time Frame: 4 years
Population: This study contains only one group. All patients received AVJ-514 device - MitraClip NT System.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Death | 5
  Stroke | 1
  Myocardial Infarction | 0
  Renal Failure | 2
  Non-elective Cardiovascular Surgery for device or procedure related Adverse Event | 0

160. Secondary Outcome: Freedom From the Components of the Primary Safety Composite of MAE
Description: as for outcome 157
Time Frame: 5 years
Reporting Status: Not Posted

161. Secondary Outcome: Number of Patients With New York Heart Association (NYHA) Functional Class
Description: Class I: Patients with cardiac disease but without resulting limitations of physical activity. Class II: Patients with cardiac disease resulting in slight limitation of physical activity. Patients are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain. Class III: Patients with cardiac disease resulting in marked limitation of physical activity. Patients are comfortable at rest. Less than ordinary physical activity causes fatigue, palpitation dyspnea, or anginal pain. Class IV: Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of cardiac insufficiency or of the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Class I | 0
  Class II | 19
  Class III | 10
  Class IV | 1

162. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: as for outcome 161
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Class I | 21
  Class II | 8
  Class III | 1
  Class IV | 0

163. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: as for outcome 161
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
Participants
  Class I | 19
  Class II | 8
  Class III | 2
  Class IV | 0

164. Secondary Outcome: Number of Participants With NYHA Functional Class
Description: as for outcome 161
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
Participants
  Class I | 18
  Class II | 8
  Class III | 2
  Class IV | 0

165. Secondary Outcome: NYHA Functional Class
Description: as for outcome 161
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
Participants
  NYHA Class I | 16
  NYHA Class II | 10
  NYHA Class III | 2
  NYHA Class IV | 0

166. Secondary Outcome: NYHA Functional Class
Description: as for outcome 161
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 24
Participants
  NYHA Class I | 15
  NYHA Class II | 9
  NYHA Class III | 0
  NYHA Class IV | 0

167. Secondary Outcome: NYHA Functional Class
Description: as for outcome 161
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 22
Participants
  NYHA I | 10
  NYHA II | 10
  NYHA III | 0
  NYHA IV | 1
  Not Available | 1

168. Secondary Outcome: NYHA Functional Class
Description: as for outcome 161
Time Frame: 5 years
Reporting Status: Not Posted

169. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire Quality of Life (KCCQ QoL) Scores
Description: KCCQ is a self-administered questionnaire that quantifies physical limitations, symptoms, self-efficacy, social interference and quality of life. This questionnaire is a reliable and responsive health status measure used in various cardiovascular research studies. A minimum mean group difference in KCCQ score of ≥5 is considered to be clinically significant. Each question responses are coded sequentially (1, 2, 3, 4, 5 and 6) from worst to best status. Scores are generated by adding points for all questions and scaled from 0 to 100, with 0 denoting the worst and 100 the best possible status.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
units on a scale | 71.8 (14.9)

170. Secondary Outcome: KCCQ QoL Scores
Description: as for outcome 169
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
units on a scale | 81.3 (17.1)

171. Secondary Outcome: KCCQ QoL Scores
Description: as for outcome 169
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
units on a scale | 79.3 (18.7)

172. Secondary Outcome: KCCQ QoL Scores
Description: as for outcome 169
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
units on a scale | 79.6 (20.5)

173. Secondary Outcome: Change in KCCQ QoL Scores From Baseline to 1 Year
Description: as for outcome 169
Time Frame: Baseline to 1 Year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
units on a scale | 6.7 (13.5)

174. Secondary Outcome: KCCQ QoL Scores
Description: as for outcome 169
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 26
score on a scale | 80.1 (17.4)

175. Secondary Outcome: KCCQ QoL Scores
Description: The Kansas City Cardiomyopathy Questionnaire is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life.
Time Frame: 3 years
Reporting Status: Not Posted

176. Secondary Outcome: KCCQ QoL Scores
Description: as for outcome 175
Time Frame: 4 years
Reporting Status: Not Posted

177. Secondary Outcome: KCCQ QoL Scores
Description: as for outcome 175
Time Frame: 5 years
Reporting Status: Not Posted

178. Secondary Outcome: SF-36 QoL Scores
Description: The Short Form(SF) (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The physical & mental functions were assessed by the Physical Component Summary (PCS) score & Mental Component Summary (MCS) score. Normal PCS and MCS scores vary depending on the demographics of the population studied. The PCS&MCS norms for 65-75 year old are 44 & 52, respectively while the norms for congestive heart failure (CHF) population are 31 & 46, respectively.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
units on a scale
  Physical Component Summary | 32.2 (15.1)
  Mental Component Summary | 53.0 (9.3)

179. Secondary Outcome: SF-36 QoL Scores
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
  The physical & mental functions were assessed by the Physical Component Summary (PCS) score & Mental Component Summary (MCS) score. Normal PCS and MCS scores vary depending on the demographics of the population studied. The PCS&MCS norms for 65-75 year old are 44 & 52, respectively while the norms for CHF population are 31 & 46, respectively.
Time Frame: 30 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
units on a scale
  Physical Component Summary | 37.5 (12.8)
  Mental Component Summary | 54.9 (7.6)

180. Secondary Outcome: SF-36 QoL Scores
Description: The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
units on a scale
  Physical Component Summary | 37.6 (17.1)
  Mental Component Summary | 53.8 (8.9)

181. Secondary Outcome: SF-36 QoL Scores
Description: as for outcome 180
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 27
units on a scale
  Physical Component Summary | 36.3 (15.3)
  Mental Component Summary | 53.1 (9.8)

182. Secondary Outcome: Change in SF-36 QoL Scores From Baseline to 1 Year
Time Frame: From baseline to 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 27
units on a scale
  Physical Component Summary | 3.7 (12.5)
  Mental Component Summary | 1.4 (8.5)

183. Secondary Outcome: SF-36 QoL Scores
Description: as for outcome 180
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 26
score on a scale
  Physical Function (PF) | 34.5 (15.8)
  Role Physical (RP) | 39.5 (12.7)
  Bodily Pain (BP) | 48.8 (12.7)
  General Health (GH) | 45.3 (8.8)

184. Secondary Outcome: Change in SF-36 QoL Scores From Baseline
Time Frame: At 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AVJ-514
Number analyzed (Participants) | 26
score on a scale
  Physical Function (PF) | 0.7 (12.4)
  Role Physical (RP) | 4.7 (14.5)
  Bodily Pain (BP) | 0.7 (13.3)
  General Health (GH) | 2.0 (8.7)

185. Secondary Outcome: Number of Participants Undergoing Mitral Valve Surgery
Time Frame: Through 5 years
Reporting Status: Not Posted

186. Secondary Outcome: Number of Participants With Additional Mitra Clip Device Intervention
Time Frame: Through 5 years
Reporting Status: Not Posted

187. Secondary Outcome: Six Minute Walk Test (6MWT) Distance
Description: The 6MWT is a practical simple test that requires a 100-ft hallway but no exercise equipment or advanced training for technicians. This test measures the distance that a patient can quickly walk on a flat, hard surface in a period of 6 minutes (the 6MWD). It evaluates the global and integrated responses of all the systems involved during exercise, including the pulmonary and cardiovascular systems, systemic circulation, peripheral circulation, blood, neuromuscular units, and muscle metabolism. It does not provide specific information on the function of each of the different organs and systems involved in exercise or the mechanism of exercise limitation, as is possible with maximal cardiopulmonary exercise testing. The self-paced 6MWT assesses the submaximal level of functional capacity.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
meters | 349.4 (118.4)

188. Secondary Outcome: Six Minute Walk Test (6MWT) Distance
Description: as for outcome 187
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
meters | 338.6 (106.5)

189. Secondary Outcome: Six Minute Walk Test (6MWT) Distance
Description: as for outcome 187
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
meters | 359.0 (111.3)

190. Secondary Outcome: Changes in Six Minute Walk Test (6MWT) Distance From Baseline to 1 Year
Time Frame: Baseline to 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
meters | 1.4 (79.1)

191. Secondary Outcome: Six Minute Walk Test (6MWT) Distance
Description: as for outcome 187
Time Frame: 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
meters | 313.7 (136.7)

192. Secondary Outcome: Changes in Six Minute Walk Test (6MWT) Distance From Baseline
Time Frame: At 24 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 25
meters | -40.8 (86.9)

193. Secondary Outcome: Six Minute Walk Test (6MWT) Distance
Description: as for outcome 187
Time Frame: 3 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 21
meters | 336.8 (119.4)

194. Secondary Outcome: Six Minute Walk Test (6MWT) Distance
Description: as for outcome 187
Time Frame: 4 years
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: Meters
Arm/Group | AVJ-514
Number analyzed (Participants) | 16
Meters | 324.3 (112.7)

195. Secondary Outcome: Six Minute Walk Test (6MWT) Distance
Description: as for outcome 187
Time Frame: 5 years
Reporting Status: Not Posted

196. Secondary Outcome: Number of Participants With Mitral Valve Surgery
Description: Surgical access to repair or replace the mitral valve. Measured per occurrence.
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

197. Secondary Outcome: Number of Participants With Mitral Valve Surgery
Description: Surgical access to repair or replace the mitral valve. Measured per occurrence.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

198. Secondary Outcome: Number of Participants With Additional AVJ-514 Device Intervention
Description: Number of participants with any additional AVJ-514 procedure after the index procedure. Measured per occurrence.
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

199. Secondary Outcome: Number of Participants With Additional AVJ-514 Device Intervention
Description: Number of participants with any additional AVJ-514 procedure after the index procedure. Measured per occurrence.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

200. Secondary Outcome: Number of Hospitalizations and Reason for Hospitalization
Time Frame: 1 year post index procedure
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 10
Participants
  Heart failure | 4
  Cardiovascular | 2
  Non-cardiovascular | 9

201. Secondary Outcome: Number of Hospitalizations
Time Frame: 24 months
Reporting Status: Not Posted

202. Secondary Outcome: Number of Hospitalizations
Time Frame: 3 years
Reporting Status: Not Posted

203. Secondary Outcome: Number of Hospitalizations
Time Frame: 4 years
Reporting Status: Not Posted

204. Secondary Outcome: Number of Hospitalizations
Time Frame: 5 years
Reporting Status: Not Posted

205. Secondary Outcome: Number of Participants With Mitral Stenosis
Description: Defined as a mitral valve orifice of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

206. Secondary Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice of less than 1.5 cm2 as measured by the site.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

207. Secondary Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

208. Secondary Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory.
Time Frame: 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

209. Secondary Outcome: Mitral Stenosis
Description: Defined as a mitral valve orifice of less than 1.5 cm2 as measured by the Echocardiography Core Laboratory.
Time Frame: 5 years
Reporting Status: Not Posted

210. Secondary Outcome: Number of Participants With Clinically Significant Atrial Septal Defect (ASD) That Requires Intervention
Description: Defect ('hole') in the septum between the left and right atria; considered clinically significant if it requires percutaneous or surgical intervention (repair of ASD completed at the time of surgery for other reasons, but not as the primary reason for surgery, is not counted as ASD.)
Time Frame: 12 months
Reporting Status: Not Posted

211. Secondary Outcome: Number of Participants With Clinically Significant ASD That Requires Intervention
Description: as for outcome 210
Time Frame: 24 months
Reporting Status: Not Posted

212. Secondary Outcome: Number of Participants With Clinically Significant ASD That Requires Intervention
Description: as for outcome 210
Time Frame: 3 years
Reporting Status: Not Posted

213. Secondary Outcome: Number of Participants With Clinically Significant ASD That Requires Intervention
Description: as for outcome 210
Time Frame: 4 years
Reporting Status: Not Posted

214. Secondary Outcome: Number of Participants With Clinically Significant ASD That Requires Intervention
Description: as for outcome 210
Time Frame: 5 years
Reporting Status: Not Posted

215. Secondary Outcome: Number of Participants With Major Bleeding
Description: Major bleeding is defined as bleeding ≥ Type 3 based on a modified Bleeding Academic Research Consortium (BARC) definition.
  Type 3:
  * Type 3a (i) Overt bleeding plus hemoglobin drop of 3 to <5 g/dL* (provided hemoglobin drop is related to bleed) (ii) Any transfusion with overt bleeding
  * Type 3b (i) Overt bleeding plus hemoglobin drop ≥5 g/dL* (provided hemoglobin drop is related to bleed) (ii) Cardiac tamponade (iii) Bleeding requiring surgical intervention for control (excluding dental/nasal/skin/hemorrhoid) (iv) Bleeding requiring intravenous vasoactive agents
  * Type 3c (i) Intracranial hemorrhage (does not include microbleeds or hemorrhagic transformation, does include intraspinal) (ii) Subcategories confirmed by autopsy or imaging or lumbar puncture (iii) Intraocular bleed compromising vision
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

216. Secondary Outcome: Number of Participants With Major Bleeding
Description: as for outcome 215
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 3

217. Secondary Outcome: Number of Participants With Usage of Concomitant Cardiac Medications
Description: Number of participants with any change in type of medication from baseline to follow-up. Measured in overall counts.
Time Frame: At baseline (Within 14 days prior to the AVJ-514 procedure)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Angiotensin converting enzyme (ACE) inhibitor | 11
  Angiotensin II receptor blocker | 5
  Aldosterone receptor blocker | 3
  Beta-blocker | 24
  Diuretics | 30
  Calcium channel blocker | 9
  Anti-Platelets | 14
  Anticoagulants | 22
  Antiarrhythmics | 8
  Cardiac glycosis (Digitalis) | 4
  Statins | 17
  Other vasodilators | 9
  Other cardiac medication | 22

218. Secondary Outcome: Number of Participants With Usage of Concomitant Cardiac Medications
Description: Number of participants with any change in type of medication from baseline to follow-up. Measured in overall counts.
Time Frame: 30 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants
  Angiotensin converting enzyme (ACE) inhibitor | 11
  Angiotensin II receptor blocker | 4
  Aldosterone receptor blocker | 3
  Beta-blocker | 25
  Diuretics | 29
  Calcium channel blocker | 6
  Anti-Platelets | 16
  Anticoagulants | 21
  Antiarrhythmics | 7
  Cardiac glycosis (Digitalis) | 4
  Statins | 17
  Other vasodilators | 4
  Other cardiac medication | 3

219. Secondary Outcome: Number of Participants With Usage of Concomitant Cardiac Medications
Description: Number of participants with any change in type of medication from baseline to follow-up. Measured in overall counts.
Time Frame: 6 months
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 29
Participants
  Angiotensin converting enzyme (ACE) inhibitor | 11
  Angiotensin II receptor blocker | 4
  Aldosterone receptor blocker | 2
  Beta-blocker | 25
  Diuretics | 27
  Calcium channel blocker | 6
  Anti-Platelets | 16
  Anticoagulants | 18
  Antiarrhythmics | 5
  Cardiac glycosis (Digitalis) | 4
  Statins | 17
  Other vasodilators | 4
  Other cardiac medication | 4

220. Secondary Outcome: Number of Participants With Usage of Concomitant Cardiac Medications
Description: Number of participants with any change in type of medication from baseline to follow-up. Measured in overall counts.
Time Frame: 1 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 28
Participants
  Angiotensin converting enzyme (ACE) inhibitor | 12
  Angiotensin II receptor blocker | 5
  Aldosterone receptor blocker | 2
  Beta-blocker | 25
  Diuretics | 27
  Calcium channel blocker | 6
  Anti-Platelets | 15
  Anticoagulants | 17
  Antiarrhythmics | 6
  Cardiac glycosis (Digitalis) | 5
  Statins | 17
  Other vasodilators | 4
  Other cardiac medication | 4

221. Secondary Outcome: Rate of Heart Failure Hospitalizations in the 1 Year Post-AVJ-514 Procedure Compared to the 1 Year Prior
Time Frame: 1 Year Pre and Post Index Procedure
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Rate of HF Hospitalization
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Rate of HF Hospitalization
  1 year pre index procedure | 0.90 [0.62 to 1.31]
  1 year post index procedure | 0.14 [0.05 to 0.37]

222. Secondary Outcome: Number of Participants With Device Embolization Requiring Surgery
Description: Device embolization is defined as detachment of the deployed AVJ-514 device from both mitral leaflets.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

223. Secondary Outcome: Number of Participants With Device Embolization Not Requiring Surgery
Description: Device embolization is defined as detachment of the deployed AVJ-514 device from both mitral leaflets.
Time Frame: 1 year
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | AVJ-514
Number analyzed (Participants) | 30
Participants | 0

224. Secondary Outcome: Regurgitant Fraction (RF)
Description: Regurgitant fraction as determined by the site. Regurgitant fraction is defined as the regurgitant volume divided by the forward stroke volume through the regurgitant valve.
Time Frame: 2 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 15
percentage of regurgitant fraction | 28.6 (15.0)

225. Secondary Outcome: Regurgitant Fraction (RF)
Description: as for outcome 224
Time Frame: 3 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 15
percentage of regurgitant fraction | 29.8 (18.5)

226. Secondary Outcome: Regurgitant Fraction (RF)
Description: as for outcome 224
Time Frame: 4 year
Population: The number of participants analyzed includes subjects who had available follow up data at that time frame.
Measure: Mean (Standard Deviation); unit: percentage of regurgitant fraction
Arm/Group | AVJ-514
Number analyzed (Participants) | 10
percentage of regurgitant fraction | 44.7 (22.9)

ADVERSE EVENTS:
Time Frame: 4 year
Arm/Group | AVJ-514
All-Cause Mortality (participants affected / at risk) | 5/30
Serious Adverse Events (participants affected / at risk) | 27/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVJ-514 (N=30)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac Failure Chronic (Cardiac disorders) | 2 (4)
Cardiac failure (Cardiac disorders) | 8 (14)
Atrial thrombus (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Cataract (Eye disorders) | 4 (5)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1)
Sick Sinus Syndrome (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4)
Bronchitis (Infections and infestations) | 2 (2)
Bronchopneumonia (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Implant Site Infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Dementia Alzheimer's Type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Ischaemic Stroke (Nervous system disorders) | 1 (1)
Senile Dementia (Nervous system disorders) | 1 (1)
Adverse Drug Reaction (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1)
Subdural Haematoma (Injury, poisoning and procedural complications) | 1 (1)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 1 (1)
Urethral Stenosis (Renal and urinary disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tooth Extraction (Surgical and medical procedures) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Polypectomy (Surgical and medical procedures) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AVJ-514 (N=30)
Anaemia (Blood and lymphatic system disorders) | 5 (7)
Nephrogenic anaemia (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrial thrombosis (Cardiac disorders) | 2 (2)
Cardiac failure (Cardiac disorders) | 3 (3)
Cardiac failure chronic (Cardiac disorders) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Atrial Tachycardia (Cardiac disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 3 (3)
Catheter site haematoma (General disorders) | 2 (2)
Catheter site haemorrhage (General disorders) | 7 (8)
Catheter site pain (General disorders) | 3 (3)
Device lead issue (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (2)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (4)
Oesophageal infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 4 (4)
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 (1)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 2 (2)
Procedural complication (Injury, poisoning and procedural complications) | 2 (3)
Procedural headache (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 (2)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (2)
Blood creatine phosphokinase mb increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 1 (1)
Brain natriuretic peptide increased (Investigations) | 1 (1)
Cardiac enzymes increased (Investigations) | 1 (1)
Echocardiogram abnormal (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 3 (3)
Helicobacter test positive (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Inflammatory marker increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Urine viscosity abnormal (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Balance disorder (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Sedation (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 2 (2)
Renal impairment (Renal and urinary disorders) | 1 (1)
Urethral pain (Renal and urinary disorders) | 1 (1)
Urethral stenosis (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Genital erythema (Reproductive system and breast disorders) | 1 (1)
Haematospermia (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Implant Site Infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 1 (2)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dementia Alzheimer's Type (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Ischaemia Stroke (Nervous system disorders) | 1 (1)
Senile Dementia (Nervous system disorders) | 1 (1)
Sudden Hearing Loss (Ear and labyrinth disorders) | 1 (1)
Tooth Extraction (Surgical and medical procedures) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes